CLINICAL TRIAL: NCT06566937
Title: The Development and Effectiveness of E-health Videos in Improving Mental Help-seeking Intention and Behaviour Among Breast Cancer Patients
Brief Title: The Effectiveness of E-health Intervention in Improving Mental Health Outcomes Among Breast Cancer Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JEP-2024-400
Record Dates: First submitted 2024-08-12; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer; Breast Neoplasms; Depression, Anxiety; Distress, Emotional
Keywords: telemedicine; e-health; help-seeking intention; behaviour
MeSH Terms: conditions — Breast Neoplasms; Depression; Anxiety Disorders; Behavior

STUDY DESIGN:
Intervention Model Description: Intervention Group: Participants in this group will receive the e-health intervention.
  Control Group: Participants in the control group will receive standard care without the digital intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in this group will receive the e-health intervention
  Interventions: Other: E-health video
- Control (No Intervention): Participants in the control group will receive standard care and Ministry of Health pamphlets without the digital intervention

INTERVENTIONS:
Other: E-health video — Length: The video is approximately 10-15 minutes long, making it concise and easy to watch in one sitting.
  Visuals: Includes engaging visuals, such as animations, graphics, and real-life footage, to illustrate key concepts and keep viewers engaged.
  Tone: The tone is supportive, empathetic, and empowering, aiming to create a positive and encouraging atmosphere.
  Arms: Intervention

SUMMARY:
Study Purpose: The study aims to assess how effective e-health interventions are at improving mental health help-seeking intentions and behaviours among breast cancer patients.

Intervention: E-health interventions will be utilized to encourage patients to seek mental health support. These interventions are designed to be accessible and convenient, offering support and information through digital platforms.

Participants: The study will involve breast cancer patients between the ages of 18 and 65.

Key Objectives:

Primary Goal: To measure any changes in patients' intentions and actions to seek mental health support before and after using e-health interventions.

Secondary Goals: To explore how these interventions impact mental health literacy, reduce self-stigma, and identify barriers and facilitators to seeking help.

Comparison: The study will compare outcomes for patients using e-health tools against those receiving traditional care without digital interventions.

Expected Outcomes: Researchers anticipate that e-health interventions will improve mental health help-seeking behaviours, enhance understanding of mental health issues, and reduce the stigma associated with seeking support.

Significance: This study could demonstrate the potential of digital health tools to support mental well-being among breast cancer patients, providing new ways to access care and overcome traditional barriers to seeking mental health support.

DETAILED DESCRIPTION:
Study Objective: The study seeks to explore how digital health interventions can enhance the willingness and actions of breast cancer patients to seek mental health support. With the rise of digital technology, there is a growing interest in how these tools can bridge gaps in healthcare access and provide timely support.

Context and Background: Breast cancer patients often face significant emotional and psychological challenges, which can affect their overall well-being and treatment outcomes. Traditional mental health services may not always be accessible due to physical, geographic, or psychological barriers. E-health interventions present an innovative solution by offering support through digital platforms that patients can access from the comfort of their homes.

Digital Interventions: These tools are designed to provide information, support, and motivation, encouraging patients to engage in mental health services.

Methodology:

Participants: The study will recruit breast cancer patients aged 18 to 65, providing a diverse representation of those affected by the condition.

Implementation: Participants will use digital interventions over a specified period, with regular assessments to monitor changes in their mental health help-seeking behaviours and intentions.

Data Collection: Researchers will track metrics such as changes in self-reported mental health literacy, attitudes toward seeking help, self-stigma on seeking help and mental help-seeking intention score.

Comparative Analysis: The study will include a control group receiving standard care without digital interventions to compare outcomes and measure the effectiveness of e-health tools.

Anticipated Benefits:

Accessibility: E-health tools can offer immediate access to resources and support, overcoming barriers such as distance and mobility.

Personalization: Digital platforms can tailor content and support to meet individual needs, enhancing engagement and effectiveness.

Empowerment: By providing information and resources, e-health interventions can empower patients to take proactive steps in managing their mental health.

Significance: The findings from this study could have significant implications for healthcare delivery, demonstrating the value of integrating digital solutions into patient care. Successful implementation of e-health interventions could lead to widespread adoption, improving mental health outcomes for breast cancer patients and potentially other patient groups facing similar challenges.

Conclusion: By leveraging the power of digital technology, this study aims to transform the landscape of mental health support for breast cancer patients, offering new pathways to care that is accessible, effective, and patient-centred.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients from all stages of the disease who are currently undergoing treatment at Institut Kanser Negara (IKN)
* Age 18 years and above
* Patients willing to participate
* Patients understand either Malay or English language

Exclusion Criteria:

* Patients with breast cancer and metastasis to the brain
* Patients who are diagnosed with mental illness
* Patients with performance status 3 and above (based on The Eastern Cooperative Oncology Group (ECOG) Scale of Performance Status)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Mental Help-Seeking Intention | baseline, 4 weeks and 12 weeks post intervention
  Help-Seeking Intention: The likelihood or willingness of breast cancer patients to seek professional mental health services.
  The mental help-seeking intention will be assessed using the Theory of Planned Behaviour (TPB) questionnaires. The help-seeking intention will be measured on a 3-item scale. Responses will be rated on a 6-point Likert scale, with higher scores indicating higher levels of help-seeking intention.
Mental Help-Seeking Behaviour | baseline, 4 weeks and 12 weeks post intervention
  The actual actions participants took to seek mental health services, such as contacting a mental health professional or accessing online resources.
  Mental help-seeking behaviour will be assessed by their behaviour of seeking or not seeking help, the answer will be yes or no

SECONDARY OUTCOMES:
Mental Health Literacy | baseline, 4 weeks and 12 weeks post intervention
  Mental health literacy refers to the knowledge and beliefs about mental disorders that aid in their recognition, management, and prevention. Evaluation: Mental Health Literacy Scale (MHLS)
Attitude of Seeking Help, Subjective Norms, Perceived Behavioural Control (PBC) | baseline, 4 weeks and 12 weeks post intervention
  Attitude towards help-seeking, subjective norms, as well as PBC, will be assessed using the TPB questionnaires
  Perceived behavioural control - PBC will be measured on a 3-item scale. Responses will be rated on a 6-point Likert scale, with higher scores indicating higher levels of behavioural control
  Subjective norms - The subjective norm will be measured on a 3-item scale. Responses will be rated on a 6-point Likert scale, with higher scores indicating higher levels of subjective norm.
  Attitude towards help-seeking - This aspect will be assessed using 5 items, which will then be evaluated on a 6-point semantic differential scale, where higher scores denote a more favourable attitude towards help-seeking.
Self-stigma of seeking help | baseline, 4 weeks and 12 weeks post intervention
  Self-stigma refers to the internalized negative perceptions and shame associated with seeking mental health support. Self-stigma in seeking help will be assessed using the Self-Stigma of Seeking Help (SSOSH) questionnaire
Anxiety and Depression | baseline, 4 weeks and 12 weeks post intervention
  The level of anxiety and depression will be measured using the Hospital Anxiety and Depression Scale (HADS). HADS is a self-reported questionnaire designed to screen anxiety and depressive in a hospital setting

CONTACTS AND LOCATIONS:
Overall Officials: Azmawati Mohammed Nawi, Principal Investigator — The National University of Malaysia
Locations (1):
- Institut Kanser Negara, Putrajaya, Malaysia

IPD SHARING:
Plan to Share IPD: No